CLINICAL TRIAL: NCT05445791
Title: Effect of Metformin Plus Tyrosine Kinase Inhibitors Compared With Tyrosine Kinase Inhibitors Alone for Patients With Advanced Non-small Cell Lung Cancer and EGFR Mutations: Phase 3 Randomized Clinical Trial
Brief Title: Metformin Plus Tyrosine Kinase Inhibitors for Treatment of Patients With Non-small Cell Lung Cancer With EGFR Mutations
Acronym: METLUNG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Coordinator of the Thoracic Oncology Unit, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: (020/023/ICI) (CEI/1421/19)
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients randomized to this study arm will be treated with tyrosine kinase inhibitors (Gefitinib 250 mg/day; afatinib 30-40 mg/day; erlotinib 150 mg/day) plus placebo 500 mg twice daily until disease progression.
  Interventions: Other: Placebo
- Metformin (Experimental): Patients randomized to this study arm will be treated with tyrosine kinase inhibitors (Gefitinib 250 mg/day; afatinib 30-40 mg/day; erlotinib 150 mg/day) plus metformin 500 mg twice daily until disease progression.
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Metformin 500 mg twice daily until disease progression.
  Arms: Metformin
Other: Placebo — Placebo 500 mg twice daily until disease progression
  Arms: Placebo

SUMMARY:
Lung cancer represents the most frequent neoplastic disease worldwide, with an annual incidence of over 2 million cases, which represents 11.6% of all cancer diagnoses. Further, it constitutes the main cause of cancer-related deaths. Among the lung cancer types, non-small cell lung cancer represents 80-85% of cases, and the majority of patients are diagnosed with locally advanced or metastatic disease, and 5-year survival rates remain discouraging in most world regions, ranging from 8-18%.

Advances in molecular biology have led to the discovery of several molecular targets and development of targeted therapy for patients with specific molecular subtypes of NSCLC. One of the most widely studied is the epidermic growth factor receptor (EGFR), which has been long recognized as a key modulator for specific tumor cell functions, and thus it has been used in drug development strategies.

Mutations in the EGFR gene are reported in 15% of all NSCLC cases, though incidence varies widely and in Mexico up to 34% of patients present with tumors with EGFR mutations. Treatment of patients with tumors with these characteristics is based on specific tyrosine kinase inhibitors (TKIs), achieving higher objective response rates and improved progression-free survival (PFS) compared with chemotherapy-based schemes. Nonetheless, despite the initial response, most patients treated with TKIs will eventually develop resistance mechanisms and present progressive disease. Consequently, the development of novel strategies to overcome TKI resistance and improve PFS of patients with NSCLC with epidermic growth factor receptor mutations (EGFRm) is priority.

Up to 30% of patients with NSCLC present with somatic mutations in the liver kinase B1 (LKB1) gene, which acts as a tumor suppressor through inhibition of mammilian target of rapamycin (mTOR). In a study which included 24 patients with LKB1 expression who received treatment with metformin + TKIs, overall survival was improved significantly, and therefore it is important to evaluate LKB1 expression in addition to mutations which could be related with treatment response in patients given metformin plus antineoplastic agents. LKB1 can activate AMP-activated protein kinase (AMPK) signaling through specific phosphorylations at aminoacid residues. AMPK can regulate cell cycle, cell proliferation and cell survival in NSCLC. Recently, the loss of expression of LKB1 has been associated with a reduced activation in AMPK using in vivo models, and increase in tumor necrosis after treatment with bevacizumab. The expression of AMPK has also been evaluated in NSCLC, a study which included 99 samples concluded that increased AMPK expression was associated with worse overall survival. Nonetheless, the association between AMPK expression and metformin treatment has not been ascertained.

Metformin is a biguanide used as treatment for type 2 diabetes. Additionally, several studies have identified a reduced incidence and mortality from diverse neoplasms in patients treated with metformin. In vitro studies have shown that metformin is cytotoxic in lung adenocarcinoma cells, producing a cell cycle arrest at G0 and G1, and it inhibits resistance to TKIs induced by Epithelial-Mesenchymal transition (EMT). Retrospective trials have also provided evidence as to the benefit of metformin in patients undergoing treatment for NSCLC. Several prospective trials have evaluated the concurrent use of metformin plus TKIs for patients with lung adenocarcinoma, though results have been controversial.

This randomized, phase 3 study will evaluate the PFS in patients with NSCLC with EGFR mutations undergoing treatment with TKIs plus placebo vs. TKIs plus metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologically confirmed diagnosis of non-small cell lung cancer (stage IIIB-IV) according to the American Joint Committee on Cancer (AJCC) eight edition.
2. Measurable disease by RECIST 1.1.
3. 18 years of age or older.
4. Functional status 0-2 as assessed by Eastern Cooperative Oncology Group (ECOG) scale.
5. Life expectancy of minimum12 weeks.
6. Patients with non-small cell lung cancer and a documented EGFR sensitizing mutation.
7. Patients without previous EGFR-TKI treatment. Previous use of chemotherapy is allowed with a washout period of at least 6 months.
8. Patients with asymptomatic brain metastases, or if symptoms are present treatment with radiotherapy (whole brain radiotherapy, stereotactic radiosurgery) or surgery must be administered.
9. Neutrophil count ≥1.5 x 103/mm3, and platelet count >100 x (103/mm3).
10. Serum bilirubin ≤1.5 the superior upper limit.
11. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2 superior upper limit (or ≤ 5 times the superior upper limit in patients with liver metastases).
12. Serum creatinine ≤ 1.5 superior upper limit, or creatinine clearance ≥ 60ml/min.
13. Full ability to complete all study procedures and follow up.
14. Women with child-bearing potential must have a negative pregnancy test within 72 hours of treatment start.
15. Patients with reproductive potential must use effective contraception.
16. Signed informed consent for participation in the study.
17. Availability of tumor tissue (pre-treatment biopsy) to determine LKB1 and AMPK status.

Exclusion Criteria:

1. Any unstable systemic disease (including active infection, grade 4 hypertension, unstable angina, congestive heart disease, hepatic diseases, renal diseases).
2. Patients previously treated with an EGFR-TKI.
3. Patients diagnosed with any other neoplastic disease in the previous 5 years (except in situ cervical carcinoma or basocellular skin cancer, treated accordingly).
4. Patients unable to receive oral medication, who require IV nourishment, or who underwent surgical procedures with affect nutrient absorption, or with an active peptic ulcer.
5. Pregnant or lactating women.
6. Patients diagnosed with type 2 diabetes or a glycated hemoglobin ≥ 6.5%.
7. Patients being currently treated with metformin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2024-07-14 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 48 months
  Time from treatment start until documented disease progression (according to RECIST criteria) or death by any cause.

SECONDARY OUTCOMES:
Overall survival | 48 months
  Time from treatment start until death by any cause.
Overall Response Rate | 3 months
  The sum of complete and partial response as assessed by RECIST criteria version 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No